CLINICAL TRIAL: NCT04502537
Title: A Prospective Cohort Study of Roxadustat for Anemia in Patients With Chronic Kidney Disease
Brief Title: Roxadustat for Anemia in Patients With CKD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20203357012
Record Dates: First submitted 2020-08-03; First posted 2020-08-06 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-10

CONDITIONS: Anemia of Chronic Kidney Disease
MeSH Terms: interventions — roxadustat; Erythropoietin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Roxadustat: treatment with roxadustat
  Interventions: Drug: Roxadustat
- erythropoietin: treatment with erythropoietin
  Interventions: Drug: erythropoietin

INTERVENTIONS:
Drug: Roxadustat — Oral
  Other Names: Roxadustat capsules
  Groups: Roxadustat
Drug: erythropoietin — injection
  Other Names: Recombinant Human Erythropoietin Injection(CHO cell)
  Groups: erythropoietin

SUMMARY:
A number of RCT studies have shown the safety and effectiveness of oral Roxadustat in the treatment of renal anemia, but there is a lack of evidence from cohort studies. A prospective cohort study is planed to conduct to evaluate the efficacy and safety of Roxadustat for renal anemia in the real world.

DETAILED DESCRIPTION:
The prevalence of anemia in patients with chronic kidney disease (CKD) (15.4%) is twice that of the general population (7.6%), and the degree of anemia increases with the severity of CKD. A number of RCT studies have shown the safety and effectiveness of oral Roxadustat in the treatment of renal anemia, but there is a lack of evidence from cohort studies. A prospective cohort study is planed to conduct to evaluate the efficacy and safety of Roxadustat for renal anemia in the real world. It is planned to continuously recruit patients with renal anemia in Shenzhen Second People's Hospital from October 2020 to June 2023. The treatment of anemia will be recorded (Roxadustat or erythropoietin), and the observation period is one year. Collect the patient's demographic characteristics, drug dosage, adjustment plan, hemoglobin. The main outcome indicators were: the average change in Hb from baseline to 28-52 weeks, and the Hb response rate reached during two consecutive visits; the secondary outcome indicators were: the maintenance rate of the target Hb level, iron metabolism indicators, 0 to 8 weeks of Hb level increase rate, dose adjustment and safety indicators. The generalized additive mixed model of repeated measures was used to analyze the changes and differences of outcome indicators in different groups. Expected results: In the cohort study, the effectiveness and safety of roxastat in the treatment of renal anemia, the starting dose and the adjustment plan, provide a basis for guiding the clinical safe and effective application of roxastat.

ELIGIBILITY:
Inclusion Criteria:

1. the patient did not receive ESA treatment.The average Hb level of the last two (at least 7 days before the start of the study treatment and during the screening period) was <10 g/dL.

   Or patients who have received ESA:

   Patients with renal anemia who received ESA for at least 4 weeks within the approved dose range in China before the screening evaluation.
2. The average Hb level of the last two (at least 7 days before the start of the study treatment and during the screening period) >=7 g/dL and <=12.0 g/dL;
3. The expected survival time is more than 1 year;

Exclusion Criteria:

1. a history of severe, chronic, end-stage or uncontrolled autoimmune liver disease, Child Pugh score was grade C, or with active hepatitis;
2. preparing for pregnancy or pregnancy or lactation;
3. having anemia caused by any other disease other than CKD, such as thalassemia, sickle cell anemia, pure red aplastic anemia, hemolytic anemia, tumor-related anemia, chemotherapy-related anemia, and myelodysplastic syndrome;
4. malignant tumor, such as prostate cancer, breast cancer, renal cell cancer or any other malignant tumor history or diagnosed
5. .Any red blood cell infusion during the screening period;
6. The patient is known to be allergic to the active substance (Roxadustat) or any excipient of the product;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Renal anemia patients who are naïve to roxadustat or ESA
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Mean value of Hb levels over time | Up to Week 52
  Hb will be measured throughout the period.
Achievement rate for target Hb level | Up to Week 52
  Percent of participants who achieved target Hb level (≥10.0 ).

SECONDARY OUTCOMES:
Mean Hb levels at 4 weeks after using roxadustat | At Week 4
  Hb levels at 4 weeks after using roxadustat
Mean Hb levels at 8 weeks after using roxadustat | At Week 8
  Hb levels at 8 weeks after using roxadustat
the dose of Roxadustat used | Up to Week 52
  the dose of Roxadustat used recorded monthly
Change from baseline in Hemoglobin (Hb) levels | Up to Week 52
  Change from baseline in Hemoglobin (Hb) levels was recorded monthly
the proportion of patients with different Hb levels | Up to Week 52
  the proportion of patients with different Hb levels
The proportion of patients with low response to ESA | Up to Week 52
  The proportion of patients with low response to ESA
Concentration of Serum iron | Up to Week 52
  Serum iron will be measured throughout the period.
Number of Participants with adverse events | Up to Week 52
  adverse events will be record throughout the period.

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Cheng, Dr., Principal Investigator — Shenzhen Second People's Hospital
Locations (1):
- Shenzhen Second People's Hospital, Shenzhen, China

IPD SHARING:
Plan to Share IPD: Undecided